CLINICAL TRIAL: NCT03904732
Title: Predictive Modelling of the Effects of Regular Low-dose Aspirin on COlorectal Cancer, Cardiovascular Disease and Safety Outcomes in Europe: PEACOCS Model EU
Brief Title: Study to Develop a Prediction Model to Understand the Effect of Low-dose Aspirin on Cancer That Develops in the Colon and/or the Rectum, Diseases That Affects the Heart or Blood Vessels and Safety Outcomes in European Countries. The Study is Also Called PEACOS Model EU
Acronym: PEACOCS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20751
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer; Cardiovascular Disease; Bleeding
MeSH Terms: conditions — Colorectal Neoplasms; Cardiovascular Diseases; Hemorrhage | interventions — Aspirin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Cohort 1: hypothetical UK populations of adults aged 50-59 take low-dose aspirin for primary prevention
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Cohort 2: hypothetical UK populations of adults aged 50-59 take low-dose aspirin for secondary prevention
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Cohort 3: hypothetical UK populations of adults aged 50-59 do not take low-dose aspirin for primary prevention
- Cohort 4: hypothetical UK populations of adults aged 50-59 do not take low-dose aspirin for secondary prevention
- Cohort 5: hypothetical UK populations of adults aged 60-69 take low-dose aspirin for primary prevention
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Cohort 6: hypothetical UK populations of adults aged 60-69 take low-dose aspirin for secondary prevention
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Cohort 7: hypothetical UK populations of adults aged 60-69 do not take low-dose aspirin for primary prevention
- Cohort 8: hypothetical UK populations of adults aged 60-69 do not take low-dose aspirin for secondary prevention

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — Low-dose acetylsalicylic acid, Aspirin (75-150 mg)
  Groups: Cohort 1; Cohort 2; Cohort 5; Cohort 6

SUMMARY:
In this study researchers want to learn more about the effect of low-dose Aspirin on cancer that develops in the colon (the longest part of the large intestine) and/or the rectum (the last several inches of the large intestine before the anus), diseases that affects the heart or blood vessels and safety outcomes. Study will focus on two groups of adults aged 50-59 and 60-69 years having an increased risk of heart and/or blood vessel disease who are taking either low-dose aspirin or no low-dose aspirin for heart and/or blood vessel disease prevention. The model will be based on information publicly available either on government organization websites or in scientific journals. Based on these data researchers will focus in a first step to build a model of 2 million adults (1 million for each age group) for the UK population and in a second step, the model will be modified for use with other European countries, to reflect the epidemiology and guidelines for aspirin use in these countries.

DETAILED DESCRIPTION:
Observational Study Model is selected as "Other" - Reason: Individual-level state transition model simulating the number of events of CRC, CVD, safety events and deaths in hypothetical cohorts of 1 million adults aged 50-59 years and 1 million adults aged 60-69 years followed for 20 years or till death, whichever comes first. The hypothetical cohorts are reflective of a population eligible for taking aspirin for primary or secondary CVD prevention.

Time Perspective is also selected as "Other"

- Reason: Individual-level state transition model built mimicking the UK population using data published in scientific international peer-reviewed journals or published data from government agencies. In a second phase, the model results will be extrapolated to other EU countries, modifying the model parameters to reflect the other EU countries epidemiology.

ELIGIBILITY:
Inclusion Criteria:

- European populations (UK and other European countries) of adults aged 50-59 and 60-69 years eligible for using aspirin for primary or secondary CVD prevention. Subjects are eligible when they have no contra-indications, and are at increased risk of CVD (primary prevention) or have suffered from a previous CVD event

Exclusion Criteria:

- None

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disease prediction model using hypothetical populations of adults aged 50-59 and 60-69 years at increased CVD (cardiovascular disease) risk, taking aspirin for CVD (primary or secondary) prevention.
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Number of myocardial infarction and ischaemic stroke | Up to 20 years
  Calculated results using a mimicked population
Number of death due to myocardial infarction or due to ischaemic stroke | Up to 20 years
  Calculated results using a mimicked population
Number of colorectal cancer (CRC) | Up to 20 years
  Calculated results using a mimicked population
Number of death due to CRC | Up to 20 years
  Calculated results using a mimicked population
Number of severe gastrointestinal (GI) bleeding requiring hospitalization | Up to 20 years
  Calculated results using a mimicked population
Number of intracranial hemorrhage (ICH) | Up to 20 years
  Calculated results using a mimicked population
Number of symptomatic peptic ulcers requiring hospitalization | Up to 20 years
  Calculated results using a mimicked population
Number of deaths due to any other cause | Up to 20 years
  Calculated results using a mimicked population

CONTACTS AND LOCATIONS:
Locations (1):
- Mimicked Population, Mimicked Population, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.